CLINICAL TRIAL: NCT01416233
Title: Autologous Fat Augmentation of Orbital Volume Using a Closed Cannula Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox, Donald Munro, M.D., P.C. (Individual)
Responsible Party: Principal Investigator, Donald M Fox, MD, Fox, Donald Munro, M.D., Fox, Donald Munro, M.D., P.C.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10.27
Record Dates: First submitted 2011-05-30; First posted 2011-08-12 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Orbital Fat Atrophy
Keywords: autologous; fat; orbit; atrophy; cannula
MeSH Terms: conditions — Platelet Glycoprotein IV Deficiency; Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- autologous fat grafting (Experimental): There is one arm of this study. People with anophthalmic sockets and orbital atrophy are given a single session of autologous fat grafting by a closed cannula technique and are observed to measure, by MRI, the amount of fat retained at one year
  Interventions: Procedure: autologous fat grafting to the orbit

INTERVENTIONS:
Procedure: autologous fat grafting to the orbit — subjects will undergo fat harvesting followed by autologous fat grafting into the orbit into their anophthalmic orbit

SUMMARY:
After enucleation or evisceration with placement of a dermis fat graft or integrated orbital implant as a primary procedure, there can be secondary loss of orbital fat volume causing regression of periocular tissue and malpositioning of the cosmetic shell. Current techniques for correction require open surgery to place a sheet/block of biocompatible material or a macroaggregate of fat into the orbit to augment orbital volume for permanent correction. Alternatively, hyaluronic acid-base fillers (Restylane, Radiesse) have been injected, but these have proved to be temporary. The current study seeks to show that a permanent augmentation of orbital volume can be achieved using a closed cannula injection of autologous fat.

DETAILED DESCRIPTION:
To date, 5 subjects have completed fat injections and 4/5 have acquired complete sets of 3 MRIs each. Data analysis has begun. The study has been extended to include 5 more subjects (total 10) to increase the number of data for analysis.

To date, the protocol has been expanded to include 10 subjects of which 6/10 have completed fat injections. The study period has been extended to include MRIs at 2 and 5 years after injection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have developed secondary orbital fat atrophy after enucleation/evisceration with or without dermis fat grafting
* standard sphere or integrated orbital implantation
* phthisis bulbi are candidates

Exclusion Criteria:

* class 3 or greater anesthesia risk
* infection
* inability to follow study protocol

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-09; Primary Completion 2017-12-10 (Actual); Study Completion 2017-12-10 (Actual)

PRIMARY OUTCOMES:
Autologous Augmentation of Orbital Volume Using a Closed Cannula Technique | 1-5 years
  Autologous fat will be injected into the orbits of anophthalmic human subjects with secondary loss of orbital volume

CONTACTS AND LOCATIONS:
Locations (1):
- New York Eye and Ear Infirmary, New York, New York, United States

REFERENCES:
- See also: further information — http://www.newyorkfami.com